CLINICAL TRIAL: NCT05849636
Title: Alerta Cannabis: Evaluación de Una Intervención a Medida Basada en el Ordenador Para la Prevención Del Consumo de Cannabis en Adolescentes de 14 a 18 Años
Brief Title: Alerta Cannabis: Evaluation of Web-based Tailored Intervention
Acronym: NOTCANNABIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Seville (Other)
Collaborators: Ministerio de Ciencia, Innovación y Universidades (Unknown); Maastricht University (Other)
Responsible Party: Principal Investigator, Marta Lima-Serrano, PhD, Associate Professor, University of Seville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PID2019-107229RA-I00
Record Dates: First submitted 2023-03-16; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Cannabis Use; Adolescent Behavior; E-health
Keywords: adolescence; cannabis use; i-change model; web-based interventions; e-health; prevention
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: A Cluster Randomized Controlled Trial is conducted to test the effectiveness of ALERTA CANNABIS in students aged 14 to 18 years. The study Will be carried out in 34 high schools from Andalusia (southern Spain), which will be randomized either to the experimental or the control condition (EC and CC). The EC will receive the ALERTA CANNABIS intervention, which consists of four sessions at school.The CC just completes the baseline and the evaluation questionnaires.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALERTA CANNABIS (Experimental): The Experimental Group receives the ALERTA CANNABIS intervention, which consists of four sessions at school (baseline questionnaire, two sessions in three scenarios: at home, celebrations, and public places, and a final evaluation). The adolescents are provided with answers related to their views of each scenario; this information is used to provide highly specific feedback regarding their knowledge, risk perception, self-esteem, attitude, social influence (modelling, norms and social pressure), self-efficacy and action plans. The post-tests will be carried out at six and twelve months from the baseline.
  Interventions: Behavioral: ALERTA CANNABIS
- CONTROL (No Intervention): Control Group: The Control Group just completes the baseline and the evaluation questionnaires. Evaluation takes place after six and twelve months from baseline

INTERVENTIONS:
Behavioral: ALERTA CANNABIS — The intervention consists of preventive messages about the benefits of not consuming cannabis, reducing the positive attitudes and encouraging the negative attitudes towards cannabis use, as well as social influence and self-efficacy, by personalized feedback. Skills and action plans are encouraged to help the student to reject cannabis use. This information is presented through different tailored messages. In addition, the participants will be able to choose avatars to accompany them during the intervention. The intervention consists of a short story about the cannabis use by adolescents.The stories take place in three different scenarios (at home, at school leaving, and in public places).
  Arms: ALERTA CANNABIS

SUMMARY:
This study consists in the the design, implementation, and evaluation of the first web-based computer tailored intervention program aimed at the prevention of cannabis use in Spanish adolescents (ALERTA CANNABIS). A Cluster Randomized Controlled Trial is conducted to test the effectiveness of ALERTA CANNABIS in students aged 14 to 18 years across 34 high schools from Andalusia (southern Spain), which are randomized either to the experimental or the control condition (EC and CC).

DETAILED DESCRIPTION:
Cannabis is the third most widespread drug and the most widely used illegal drug in Spanish and Andalusian adolescents aged 14 to 18 years, representing 8 out of 10 admissions to treatment for drug dependency in minors. It is necessary to continue investing in research applied to the prevention of cannabis consumption in order to develop scientifically validated strategies that can become preventive policies. The objective of the project is to contribute to the prevention of cannabis use in children, through the development, implementation and evaluation of the cost-effectiveness of a web-based-computer-tailoring and gamified learning intervention, having as reference the integrated theoretical model on adoption of health behaviors, the I-Change model. The starting hypothesis is that the application of this program, ALERTA CANNABIS, to children from 14 to 18 years old at the school context, will be cost-effective for reducing the prevalence of cannabis use.

A cluster randomized controlled trial will be carried out, with an intervention group, which will receive the ALERTA CANNABIS intervention and a waiting list control group. The following phases will be followed: design, implementation, cost-effectiveness evaluation (at 6 and 12 months), and dissemination of results.

ALERT CANNABIS will carry out an individualized advice, by means of pre-established messages, but generated based on the characteristics detected in a questionnaire (for example, the user's first name and taking into account the gender perspective, different types of reinforcement, etc.). In addition, it will use gamification techniques (videos, incentives, rankings) to encourage motivation and adherence to the intervention. The intervention will address motivational factors associated of cannabis use such as attitude, social influences, self-efficacy and intention.

The sample will consist of 1850 Andalusian students aged 14 to 18 enrolled in public high schools of the Andalusian provinces of Seville, Cordoba, Huelva, Cádiz, Granada and Malaga, 37 class groups by condition for the cluster design. Both, for the initial study and for the evaluation of cost-effectiveness, an online questionnaire applied in the school context will be used, with the variables resulting from the prevalence of cannabis use (in life, in the last 6 months, in last month), cannabis abuse using the cannabis abuse screening test (CAST) and health-related quality of life in terms of quality-adjusted life years (QALY). Confidentiality will be ensured in accordance with Royal Decree-Law 5/2018, of July 27, on the Protection of Personal Data. Informed consent will be requested.

If the cost-effectiveness of the program is demonstrated, it can be disseminated by becoming a public health policy.

ELIGIBILITY:
Criteria: Inclusion Criteria:

* Students aged 14 to 18 years.
* Enrolled in Andalusian public high schools.
* Access to the Internet at the school and an equipped information and communication technology (ICT) room.

Exclusion Criteria:

* Language barriers.
* Previous participation in prevention programs for cannabis use.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1850 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
cannabis use lifetime | six months after the baseline
  cannabis use lifetime
cannabis use lifetime | twelve months after the baseline
  cannabis use lifetime
cannabis use last 6 months (long-term) | six months after the baseline
  cannabis use lifetime
cannabis use last 6 months (long-term) | twelve months after the baseline
  cannabis use lifetime
cannabis use last 30 days (recent use) | six months after the baseline
  cannabis use last 30 days (recent use)
cannabis use last 30 days (recent use) | twelve months after the baseline
  cannabis use last 30 days (recent use)

SECONDARY OUTCOMES:
Intention to use cannabis | six months after the baseline
  Intention to use cannabis in the future
Intention to use cannabis | twelve months after the baseline
  Intention to use cannabis in the future
Intention to change cannabis consumption | six months after the baseline
  Intention to change cannabis consumption
Intention to change cannabis consumption | twelve months after the baseline
  Intention to change cannabis consumption

CONTACTS AND LOCATIONS:
Overall Officials: Marta Lima Serrano, Principal Investigator — University of Seville
Locations (1):
- University of Sevilla, Seville, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lima-Serrano M, Barrera-Villalba C, Mac-Fadden I, Mesters I, de Vries H. Alerta Cannabis: A Tailored-Computer Web-Based Program for the Prevention of Cannabis Use in Adolescents: A Cluster-Randomized Controlled Trial Protocol. BMC Nurs. 2024 Apr 10;23(1):239. doi: 10.1186/s12912-024-01889-x. PMID 38600496